CLINICAL TRIAL: NCT04624633
Title: A Phase 2 Study of Acalabrutinib, Umbralisib, and Ublituximab (AU2) in Relapsed and Previously Untreated CLL Patients
Brief Title: Acalabrutinib, Umbralisib, and Ublituximab (AU2) In Relapsed and Untreated CLL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer R. Brown, MD, PhD (Other)
Collaborators: AstraZeneca (Industry); TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jennifer R. Brown, MD, PhD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-394
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Relapsed Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Relapsed Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; umbralisib; ublituximab; LFB-R603

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1-Relapsed Disease (Experimental): Participants with relapsed disease
  * Treatment with Acalabrutinib & Umbralisib beginning C1D1,
  * Ublituximab beginning C7D1
  * Assessment of treatment response
  * Treatment continues for a maximum of 24 cycles. Participants followed post treatment for a maximum of 5 years
  Interventions: Drug: Acalabrutinib; Drug: Umbralisib; Drug: Ublituximab
- Cohort 2-Treatment Naive (Experimental): Participants with previously untreated disease
  * Treatment with Acalabrutinib & Umbralisib beginning C1D1,
  * Ublituximab beginning C7D1
  * Assessment of treatment response
  * Treatment continues for a maximum of 24 cycles. Participants followed post treatment for a maximum of 5 years
  Interventions: Drug: Acalabrutinib; Drug: Umbralisib; Drug: Ublituximab

INTERVENTIONS:
Drug: Acalabrutinib — Oral, twice a day, predetermined dosage
  Other Names: Calquence
Drug: Umbralisib — Oral, once a day, predetermined dosage, each 28 day cycle up to 24 cycles
  Other Names: RP5264
Drug: Ublituximab — 28 day cycle, starting cycle 7 via iv, on at predetermined dosage and timepoints in each cycle
  Other Names: LFB-R603

SUMMARY:
This study is testing the effectiveness of the study drug combination of acalabrutinib, umbralisib, and ublituximab in participants with Chronic Lymphocytic leukemia (CLL).

The names of the study drugs involved in this study are/is:

* Acalabrutinib (CALQUENCE®, ACP-196)
* Umbralisib (TGR-1202)
* Ublituximab (TG-1101)

DETAILED DESCRIPTION:
In this research study, Investigators are exploring the combination of acalabrutinib, umbralisib, and ublituximab and hoping to determine if the combination is effective at controlling cancer growth in participants with CLL.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive the study drugs for a maximum of 24 cycles (2 years) and will be followed for a maximum of 5 years after discontinuing the study drugs.

The names of the study drugs involved in this study are/is:

* Acalabrutinib (CALQUENCE®, ACP-196)
* Umbralisib (TGR-1202)
* Ublituximab (TG-1101)

It is expected that about 60 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drugs to learn whether the drugs work in treating a specific disease. "Investigational" means that the drugs are being studied.

* The U.S. Food and Drug Administration (FDA) has not approved umbralisib or ublituximab as a treatment for any disease.
* The U.S. Food and Drug Administration (FDA) has approved acalabrutinib for CLL, but not in this combination.

  * Acalabrutinib is a type of drug called a kinase inhibitor. It blocks a type of protein called Bruton Tyrosine Kinase (BTK) that helps CLL cells live and grow. By blocking BTK, acalabrutinib may kill cancer cells or stop them from growing.
  * Umbralisib is an investigational drug which blocks a protein called PI3K. PI3K is a protein that helps CLL cells grow.
  * Ublituximab is a type of investigational drug called a monoclonal antibody. A monoclonal antibody is a type of protein made in the laboratory that can locate and bind to substances in the body, including tumor cells. By binding to the tumor cells, the antibody might prevent the tumor cell from growing and spreading.

As of March 2023, TG therapeutics has decided to no longer provide umbralisib, ublituximab and funding for this study. Study participants still on treatment will still have access to acalabrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) per International Workshop on CLL (iwCLL) 2018 criteria.1
* Participants must have an indication for treatment as defined by iwCLL 2018 criteria.1
* Participants must have measurable disease, defined as lymphocytosis > 5,000 / μL, or palpable or CT measurable lymphadenopathy ≥ 1.5 cm, or bone marrow involvement ≥ 30%.
* For enrollment to Cohort 1: Participants must have relapsed or refractory disease as per iwCLL 2018 criteria,1 and must have received no more than 2 prior lines of anti-cancer therapy.
* For enrollment to Cohort 2: Participants must have previously untreated disease (i.e.

must not have received any prior systemic therapy for CLL or SLL).

* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of umbralisib, acalabrutinib, and ublituximab in participants < 18 years of age and CLL is extremely rare in this population, children are excluded from this study.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%, see Appendix A).
* Participants must have adequate organ and marrow function as defined below:

  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) (unless due to hemolysis or Gilbert's disease, in which ≤ 3 × institutional ULN is acceptable)
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 × institutional ULN, OR
  * AST (SGOT) and ALT (SGPT) ≤ 5 × institutional ULN if there is hemolysis or documented disease involvement in the liver
  * Calculated creatinine clearance ≥ 30 mL/min (as calculated by the Cockcroft-Gault formula)
  * Platelet count ≥ 50,000/mcL, unless there is bone marrow involvement with disease
  * PT-INR or aPTT ≤ 2 × institutional ULN
  * Absolute neutrophil count (ANC) ≥ 750 mm3
  * Hemoglobin (Hgb) > 8 g/dL
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of umbralisib, acalabrutinib, or ublituximab on the developing human fetus are unknown. For this reason and because anti-cancer agents are known to be teratogenic, women of child-bearing potential and men must agree to use highly effective methods of contraception. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated on this protocol must agree to use highly effective contraception prior to the study, for the duration of study participation, and 4 months after completion of umbralisib, acalabrutinib, or ublituximab administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow and retain oral medication.
* Participants must be able to receive prophylactic anti-pneumocystis jiroveci pneumonia (PJP) and anti-viral therapy

Exclusion Criteria:

* Participants with progressive or refractory disease while receiving either a BTK inhibitor or PI3K inhibitor. Prior exposure to either a BTK inhibitor, PI3K inhibitor, or both is acceptable as long as the participant's disease did not progress during active therapy with the agent(s).
* Participants who have undergone a major surgical procedure within 28 days of the first dose of study drug. If a participant had major surgery greater than 28 days prior to the first dose of study drug, they must have recovered adequately from any adverse event and/or complications from the intervention prior to the first dose (as judged by the treating investigator). For enrollment to Cohort 1: receipt of prior BTK inhibitor treatment within 7 days, or any other anti-cancer therapy (e.g. chemotherapy, immunotherapy, radiation, biologic therapy or any investigational agent) within 21 days of the first dose of study drug.
* Participants who are receiving any other investigational agents.
* History of prior allogeneic stem cell transplant.
* History of autologous hematologic stem cell transplant within 6 months of the first dose of study drug.
* Participants with known Richter's transformation, or histological transformation from CLL to large cell lymphoma.
* Participants with known CNS involvement, because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with no known history of CNS leukemia are not required to undergo CT scan or lumbar puncture (LP) for trial eligibility unless the participant is symptomatic as judged by the treating investigator.
* Participants with uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP).
* Participants with active clinically significant bleeding or history of bleeding diathesis (e.g. hemophilia or von Willebrand disease).
* Participants requiring or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (other anticoagulants are permitted).
* Participants with a history of significant cerebrovascular disease/event within 6 months before the first dose of study drug, including stroke or intracranial hemorrhage.
* Participants with uncontrolled intercurrent illness, including but not limited to: unstable angina pectoris, cardiac arrhythmia, or poorly controlled and clinically significant atherosclerotic vascular disease (including patients who required angioplasty, cardiac or vascular stenting within 6 months prior to the first dose of study agent), myocardial infarction within 6 months of screening, congestive heart failure, or patients with Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Note: participants with controlled, asymptomatic atrial fibrillation are permitted to enroll on study. Concomitant use of medication known to cause QT prolongation or torsades de pointes should be used with caution and at investigator discretion.
* Individuals with a history of a different malignancy are ineligible with the following exceptions: individuals who have been treated and are disease-free for a minimum of 2 years prior to study enrollment, or individuals who are deemed by the treating investigator to be at low risk for disease recurrence. Additionally, individuals with the following cancers are eligible if diagnosed and curatively treated within the past 2 years: basal or squamous cell carcinomas of the skin, and breast or cervical carcinomas in situ.

Prostate cancer on observation, with stable PSA for 6 months, is also eligible.

* Participants who require ongoing immunosuppressive therapy including systemic corticosteroids (prednisone or equivalent ≤ 10 mg daily is permitted). Topical, inhaled, and ophthalmologic steroids are permitted.
* Participants with a history of inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis).
* Participants with irritable bowel syndrome (IBS) with greater than 3 loose stools per day at baseline.
* Participants with evidence of ongoing systemic bacterial, fungal, or viral infection, except localized fungal infections of the skin or nails. NOTE: participants may be receiving prophylactic antiviral or antibacterial therapies at the treating investigator's discretion. Use of anti-pneumocystis and antiviral prophylaxis is required.
* Participants with a known history of progressive multifocal leukoencephalopathy (PML).
* Participants with evidence of chronic active Hepatitis B (HBV, not including patients with prior hepatitis B vaccination or positive serum Hepatitis B antibody), chronic active

Hepatitis C infection (HCV), active cytomegalovirus (CMV), or known history of human immunodeficiency virus (HIV):

* If HBc antibody is positive, the subject must be evaluated for the presence of HBV DNA by PCR (see Appendix B). Subjects with positive HBc antibody and negative HBV DNA by PCR are eligible but serial monitoring of HBV DNA by PCR is required, see Section 5.4. Subjects with positive HBV DNA by PCR are not eligible.
* Participants with positive HBsAg are to be excluded.
* If HCV antibody is positive, the subject must be evaluated for the presence of HCV RNA by PCR. Subjects with positive HCV antibody and negative HCV RNA by PCR are eligible. Subjects with positive HCV RNA by PCR are not eligible.
* If the subject is CMV IgG or CMV IgM positive, the subject must be evaluated for the presence of CMV DNA by PCR. Subjects who are CMV IgG or CMV IgM positive but who are CMV DNA negative by PCR are eligible, anti-viral prophylaxis should be considered per treating investigator discretion.

  * History of allergic reactions attributed to study drugs including active product or excipients, or compounds of similar chemical or biologic composition to acalabrutinib, umbralisib, or ublituximab, including participants with a history of anaphylaxis (excluding infusion-related reactions) in association with previous anti-CD20 administration.
  * Participants requiring concomitant treatment with any medications or substances that are strong inhibitors or inducers of CYP3A4 at the time of study enrollment. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
  * Participants requiring concomitant treatment with proton pump inhibitors (e.g.omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole) at the time of study enrollment. Note: participants receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids prior to the first dose of study medication are eligible.
  * Participants with psychiatric illness/social situations that would limit compliance with study requirements.
  * Pregnant women are excluded from this study because acalabrutinib, umbralisib, and ublituximab are anti-cancer agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with acalabrutinib, umbralisib, or ublituximab, breastfeeding must be discontinued prior to the initiation of study treatment. A negative serum pregnancy test is required for women of childbearing potential within 3 days prior to Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2028-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Yin Y, Xu H, He L, Brown JR, Mato AR, Aittokallio T, Skanland SS. Protein Profiles Predict Treatment Responses to the PI3K Inhibitor Umbralisib in Patients with Chronic Lymphocytic Leukemia. Clin Cancer Res. 2025 May 15;31(10):1943-1955. doi: 10.1158/1078-0432.CCR-24-2911. PMID 40085050

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Relapsed Disease: Participants with relapsed disease
  * Treatment with Acalabrutinib & Umbralisib beginning C1D1,
  * Ublituximab beginning C7D1
  * Assessment of treatment response
  * Treatment continues for a maximum of 24 cycles. Participants followed post treatment for a maximum of 5 years
- Cohort 2 - Treatment Naive: Participants with previously untreated disease
  * Treatment with Acalabrutinib & Umbralisib beginning C1D1,
  * Ublituximab beginning C7D1
  * Assessment of treatment response
  * Treatment continues for a maximum of 24 cycles. Participants followed post treatment for a maximum of 5 years
Period: Overall Study
Arm/Group | Cohort 1 - Relapsed Disease | Cohort 2 - Treatment Naive
Started | 8 | 21
Completed | 7 | 20
Not Completed | 1 | 1
Not completed — Subject Needed Surgery, Radiation or Other Therapy | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Relapsed Disease | Cohort 2 - Treatment Naive | Total
Number analyzed (Participants) | 8 | 21 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [58 to 71] | 67 [58.75 to 75] | 63 [57 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 5 | 13 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 2 | 2
  White | 7 | 18 | 25
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate After 24 Cycles
Description: The CR Rate is defined as the proportion of participants achieving complete remission (CR) based on 2018 IW-CLL criteria.
Time Frame: According to this endpoint is after 24 cycles. Overall median number of cycles is 24 with range 1-25.
Population: Patients who completed 24 cycle of treatment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1 - Relapsed Disease | Cohort 2 - Treatment Naive
Number analyzed (Participants) | 6 | 14
proportion of participants | 0.33 [0.043 to 0.777] | 0.29 [0.084 to 0.582]

2. Secondary Outcome: Partial Remission (PR) Rate After 24 Cycles
Description: The PR Rate is defined as the proportion of participants achieving partial remission (PR) based on 2018 IW-CLL criteria.
Time Frame: According to this endpoint is after 24 cycles. Overall median number of cycles is 24 with range 1-25.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1 - Relapsed Disease | Cohort 2 - Treatment Naive
Number analyzed (Participants) | 6 | 14
proportion of participants | 0.66 [0.22 to 0.88] | 0.57 [0.29 to 0.77]

3. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last dsease assessment.
Time Frame: Disease will be evaluated through imaging at cycle 1 day 1, 8, and 15, cycle 2-6 and cycle 8-25 day 1, and cycle 7 day 1, 2 and 8. Observation on treatment up to approximately 25 cycles. In long-term follow-up, survival follow-up up to 5 years.
Reporting Status: Not Posted, anticipated posting 2028-11

ADVERSE EVENTS:
Time Frame: Adverse events (AE) will be evaluated through imaging at cycle 1 day 1, 8, and 15, cycle 2-6 and cycle 8-25 day 1, and cycle 7 day 1, 2 and 8. AE observation on treatment up to approximately 25 cycles.
Arm/Group | Cohort 1 - Relapsed Disease | Cohort 2 - Treatment Naive
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/21
Serious Adverse Events (participants affected / at risk) | 7/8 | 16/21
Other Adverse Events (participants affected / at risk) | 8/8 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Relapsed Disease (N=8) | Cohort 2 - Treatment Naive (N=21)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 5
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 4
Neutrophil count decreased (Investigations) | 5 | 6
Platelet count decreased (Investigations) | 0 | 2
Weight loss (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Relapsed Disease (N=8) | Cohort 2 - Treatment Naive (N=21)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 3 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 2
Eye disorders - Other, specify (Eye disorders) | 0 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 3
Fever (General disorders) | 2 | 1
Generalized edema (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 4 | 12
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 0 | 4
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 5
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Akathisia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Extrapyramidal disorder (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 4
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 3
Hypotension (Vascular disorders) | 2 | 2
Thromboembolic event (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04624633/Prot_SAP_000.pdf